CLINICAL TRIAL: NCT04907994
Title: Impact of Containment on Primary Care Management and Clinical Adverse Events Non-related to COVID-19 in Older Patients and/or With Chronic Diseases During the Epidemic. The COVIMEGE French Retrospective Cohort Study.
Brief Title: Containment Impact on Primary Care & Adverse Events Unrelated to COVID-19 in Older Patients and/or With Chronic Diseases
Acronym: COVIMEGE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201045
Record Dates: First submitted 2021-05-14; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: Containment; Primary care; Clinical adverse events; Older patients; Chronic diseases patients
MeSH Terms: conditions — COVID-19 | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older patients and/or with chronic diseases: Retrospective cohort study of exposed/unexposed individuals in the national health data system (SNDS). The study population is composed of individuals aged 70 years or older and patients with a chronic disease. Exposure to containment is defined as the period between 17 March 2020 (beginning of week 12, start of containment) and 10 May 2020 (end of week 19, end of containment). The end of monitoring is set at 12 months after the start of the containment, on 17 March 2021. The unexposed group consists of random samples of comparable individuals (aged 70 years or older and/or chronically ill) for the two years prior to the outbreak (2015 and 2016). The second study period (May 10, 2020 to March 17, 2021) may be subdivided depending on the evolution of the health crisis and the governmental measures adopted. Measurement of the outcome measures and comparison between exposed and unexposed will be carried out at the end of each of the two periods.
  Interventions: Other: Cohort

INTERVENTIONS:
Other: Cohort — Nothing. Only implementation of a cohort with data collection via the SNDS.

SUMMARY:
In 2017, 10.7 million people affiliated to the general health insurance scheme benefited from the "Long-term condition" scheme, i.e. 17% of insured patients. Most of these patients suffer from chronic diseases requiring regular medical and paramedical follow-up. During the first containment period of the SARS-CoV-2 epidemic, the French government's messages were to call the Urgent Medical Assistance Service (15) and not to go directly to the general practitioner (GP), favouring teleconsultations. Other countries have adopted the same strategy. Mortality rates due to SARS-CoV-2 infection were higher in elderly patients and/or those with co-morbidities, particularly heart failure, hypertension, respiratory failure and diabetes. The elderly and patients with chronic cardiometabolic and respiratory diseases should therefore be particularly protected during the epidemic. However, these populations also need close monitoring to avoid acute decompensation of their chronic diseases or loss of autonomy. However, during the first containment, general practitioners and other medical and paramedical ambulatory health professionals perceived a notable decrease in their daily activity, including for their chronic and/or elderly patients who may not have called for a visit, consultation and/or access to telemedicine. "Public Health France" also reported a decrease in consultations with GPs at the beginning of the lockdown, a decrease in the number of emergency room visits and hospitalizations for cardio and neurovascular diseases. The investigators hypothesise that under-attendance of primary care services during the epidemic is associated with excess mortality and morbidity unrelated to COVID-19.

The main objective is to assess non-COVID-19 related overmortality during the containment period and 12 months after the start of containment, in a population of elderly and/or chronically ill patients in France. The overmortality will be assessed globally and according to individual and contextual characteristics such as gender, age, place of residence, pre-existing morbidity and socio-economic level.

DETAILED DESCRIPTION:
Context and hypothesis: In 2017, 10.7 million people affiliated to the French general health insurance scheme benefited from the "Long Term Affection" scheme that waives copayments related to long-term illness, i.e. 17% of the insured patients. They are mostly patients with chronic diseases requiring a regular medical and allied health and nursing care follow-up. During the SARS-CoV-2 epidemic and containment period since March 17th 2020, the French government's messages were to call the Urgent Medical Assistance Service and not to directly visit the GP except for a teleconsultation. Other countries have adopted the same strategy. Mortality rates due to SARS-CoV-2 infection were dramatically high in older patients and/or with comorbidity. In China, the case fatality rate (CFR) was 15% in patients older than 80 and in the United States, 80% of deaths occurred among adults aged 65 years. The CFR was also high in patients with underlying comorbidities, in particular heart failure, hypertension, respiratory insufficiency and diabetes. Elderly and patients with cardio-metabolic and respiratory chronic diseases therefore needed to be particularly protected during the epidemic.

However, these populations also need close management for preventing acute decompensations of chronic diseases or loss of autonomy. During containment, GPs and other medical/allied health/nurse ambulatory health providers perceived a notable decrease in their daily practice activity, including for their chronic and/or elderly patients who may not have called for a visit and/or did not have access to telemedicine. The French Public Health Agency ("Public Health France") reported a decrease in GPs visits at the start of containment, a decrease in the number of emergency visits and in hospitalizations for cardio and neurovascular diseases.

The investigators postulate that under-attendance of primary care services during the epidemic is associated with over-mortality and morbidity non-related to COVID-19.

Main Objective: To assess over-mortality non-related to COVID-19 during the first containment for SARS-CoV-2 outbreak and at 12 months, in a population of elderly and patients with chronic conditions in France. Over-mortality will be assessed globally and according to baseline individual and contextual characteristics such as area of residence, morbidity burden or socioeconomic position.

Secondary objectives: The secondary objectives concern more specifically the effect of under-attendance of primary care services due to containment, on morbidity and mortality at the end of the 12 months follow-up.

* To measure primary care healthcare utilization during containment in this population. Utilization will be assessed through the secondary endpoints related to ambulatory care.
* To analyze the effect of ambulatory healthcare utilization during the containment on non COVID-related morbidity (through the secondary endpoints related to hospital care) and mortality at the end of follow-up

Method and population:

Experimental design: Retrospective exposed/non-exposed (1:1) cohort study in the French National Health Data System (SNDS).

Endpoints:

* The primary endpoint is non-COVID-19 related mortality.
* The secondary outcome will be the use of primary care during period 1 and will be assessed through the number of consultations, teleconsultations and visits by general practitioners, and paramedical professionals (nurses and physiotherapists).

The use of specialist doctors will also be described.

Main inclusion criteria:

The study population is composed of elderly (aged 70 or older) and adult patients with a long-term illness (ALD).

Exposition to containment is defined as the period between March 17,2020 (beginning of week 12, start of containment) and May 10, 2020 (end of week 19, end of containment). The end of follow-up is set at 12 months after the start of containment, at March 17, 2021.

The non-exposed group is composed of elderly (aged 70 or older) and patients with a long-term illness (ALD) for the 2 years before epidemic (2025-2016).

Observed cases in the exposed group will be compared to expected cases estimated among the non-exposed group, for the entire study population and in sub-groups defined upon area of residence, morbidity status and socioeconomic position.

Sample size: Considering the proportion of older patients (9%), of patients suffering from chronic disease (17%) and the overlap between age and disease prevalence, the investigator expect to include approximately 18 000 000 patients.

Information for participants: Waiver of information for participants Origin of personal health data (source used): "National Health Data System"

Expected results: To quantify over-mortality non-related to COVID-19 risk in elderly and patients with chronic conditions, in order to guide public health policy: adapt government messages, improve GP-follow-up and primary care response for a future health epidemic. To identify risk factors associated with morbimortality, in particular variation of primary care utilization in order to adapt public health policy and messages to both the population and GPs.

Study duration: 30 months

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 or older and/or identification of at least one of the chronic pathologies listed in the protocol before the start of confinement (03/17/2020, start of the 12th week of the year)
* Presence in the SNDS databases throughout the duration of the follow-up (12 months post-inclusion).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is made up of people aged 70 or over and / or suffering from chronic pathologies.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Non-COVID-19 related mortality | - Exhibition to containment (March 17, 2020 to May 10, 2020);- End of containment to end of follow-up (May 11, 2020 to March 17, 2021)
  Non-COVID-19 related mortality

SECONDARY OUTCOMES:
Healthcare utilization (Consultation, visits and teleconsultations ; drug delivery ; biological and radiological procedure). | - Exhibition to containment (March 17, 2020 to May 10, 2020);- End of containment to end of follow-up (May 11, 2020 to March 17, 2021)
  Consultations, visits and teleconsultations with a general practitioner, a specialist doctor, a nurse or allied health; drug delivery ; biological and radiological procedures.
Utilization of hospital services after containment | - End of containment to end of follow-up (May 11, 2020 to March 17, 2021)
  Hospitalizations (all-causes and non-related to COVID-19), intensive care admissions (all-causes and non-related to COVID-19) and emergency visits (causes are not available).

CONTACTS AND LOCATIONS:
Overall Officials: Florence CANOUI-POITRINE, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Emilie FERRAT, MD, PhD, Study Director — Inserm - Université Paris Est Créteil; Panayotis CONSTANTINOU, MD, PhD, Study Director — Caisse nationale de l'assurance maladie, direction de la stratégie, des études et des statistiques
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No
Datas are own by "Assistance Publique - Hôpitaux de Paris", please contact sponsor for further information.